CLINICAL TRIAL: NCT04440514
Title: Endoscopic Preperitoneal Parastomal Hernia Repair (ePauli Repair)
Acronym: ePauli
Status: Recruiting | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: 137157
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Parastomal Hernia
Keywords: hernia; parastomal; robotic; laparoscopic; transversus abdominis release; repair; incisional
MeSH Terms: conditions — Hernia; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endoscopic preperitoneal repair of parastomal hernia — repair of parastomal hernia after the Sugarbaker principle with TAR and preperitoneal mesh reinforcement
  Other Names: ePauli

SUMMARY:
Observational study on laparoscopic and robotic extraperitoneal mesh repair of parastomal hernia, employing TAR.

DETAILED DESCRIPTION:
Endoscopic trans-abdominal preperitoneal plasty (TAPP) for parastomal hernia employing transversus abdominis release component separation (TAR) and reinforcement with mesh after the Sugarbaker principle, but placing mesh extraabdominally, anteriorly to the transversalis fascia. Laparoscopic and robotic procedures. Repair of concomitant midline hernia with endoscopic enhanced-view Rives-Stoppa technique.

ELIGIBILITY:
Inclusion Criteria:

* parastomal hernia with need of repair

Exclusion Criteria:

* < 18 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with permanent ostomy and parastomal hernia in need of repair
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 month
  Per- and post-operative complications

SECONDARY OUTCOMES:
Late complications | 2 years
  Stoma function, pain, mesh complications
Recurrence of hernia | 2 years
  Hernia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: jan r lambrecht, PhD, Principal Investigator — Sykehuset Innlandet Hospital Trust
Locations (2):
- Norway (2):
  - Sykehuset Innlandet Hospital Trust, Brumunddal
  - Sykehuset Innlandet HF, Hamar

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Background] Gavigan T, Stewart T, Matthews B, Reinke C. Patients Undergoing Parastomal Hernia Repair Using the Americas Hernia Society Quality Collaborative: A Prospective Cohort Study. J Am Coll Surg. 2018 Oct;227(4):393-403.e1. doi: 10.1016/j.jamcollsurg.2018.07.658. Epub 2018 Aug 4. PMID 30081081
- [Background] Nasvall P, Rutegard J, Dahlberg M, Gunnarsson U, Strigard K. Parastomal Hernia Repair with Intraperitoneal Mesh. Surg Res Pract. 2017;2017:8597463. doi: 10.1155/2017/8597463. Epub 2017 Oct 24. PMID 29204515
- [Background] Hansson BM, Slater NJ, van der Velden AS, Groenewoud HM, Buyne OR, de Hingh IH, Bleichrodt RP. Surgical techniques for parastomal hernia repair: a systematic review of the literature. Ann Surg. 2012 Apr;255(4):685-95. doi: 10.1097/SLA.0b013e31824b44b1. PMID 22418006
- [Background] DeAsis FJ, Lapin B, Gitelis ME, Ujiki MB. Current state of laparoscopic parastomal hernia repair: A meta-analysis. World J Gastroenterol. 2015 Jul 28;21(28):8670-7. doi: 10.3748/wjg.v21.i28.8670. PMID 26229409
- [Background] Pauli EM, Juza RM, Winder JS. How I do it: novel parastomal herniorrhaphy utilizing transversus abdominis release. Hernia. 2016 Aug;20(4):547-52. doi: 10.1007/s10029-016-1489-3. Epub 2016 Mar 29. PMID 27023876
- [Background] Jones CM, Winder JS, Potochny JD, Pauli EM. Posterior Component Separation with Transversus Abdominis Release: Technique, Utility, and Outcomes in Complex Abdominal Wall Reconstruction. Plast Reconstr Surg. 2016 Feb;137(2):636-646. doi: 10.1097/01.prs.0000475778.45783.e2. PMID 26818302
- [Background] Tastaldi L, Haskins IN, Perez AJ, Prabhu AS, Rosenblatt S, Rosen MJ. Single center experience with the modified retromuscular Sugarbaker technique for parastomal hernia repair. Hernia. 2017 Dec;21(6):941-949. doi: 10.1007/s10029-017-1644-5. Epub 2017 Aug 24. PMID 28840354
- [Background] Antoniou SA, Agresta F, Garcia Alamino JM, Berger D, Berrevoet F, Brandsma HT, Bury K, Conze J, Cuccurullo D, Dietz UA, Fortelny RH, Frei-Lanter C, Hansson B, Helgstrand F, Hotouras A, Janes A, Kroese LF, Lambrecht JR, Kyle-Leinhase I, Lopez-Cano M, Maggiori L, Mandala V, Miserez M, Montgomery A, Morales-Conde S, Prudhomme M, Rautio T, Smart N, Smietanski M, Szczepkowski M, Stabilini C, Muysoms FE. European Hernia Society guidelines on prevention and treatment of parastomal hernias. Hernia. 2018 Feb;22(1):183-198. doi: 10.1007/s10029-017-1697-5. Epub 2017 Nov 13. PMID 29134456
- [Background] Belyansky I, Reza Zahiri H, Sanford Z, Weltz AS, Park A. Early operative outcomes of endoscopic (eTEP access) robotic-assisted retromuscular abdominal wall hernia repair. Hernia. 2018 Oct;22(5):837-847. doi: 10.1007/s10029-018-1795-z. Epub 2018 Jul 4. PMID 29974283
- [Background] Imamura K, Takada M, Umemoto K, Furukawa S, Ambo Y, Nakamura F. Laparoscopic parastomal herniorrhaphy utilizing transversus abdominis release and a modified Sugarbaker technique: A case report. Asian J Endosc Surg. 2021 Jan;14(1):106-108. doi: 10.1111/ases.12804. Epub 2020 Jun 3. PMID 32495518
- [Background] Zolin SJ, Fafaj A, Krpata DM. Transversus abdominis release (TAR): what are the real indications and where is the limit? Hernia. 2020 Apr;24(2):333-340. doi: 10.1007/s10029-020-02150-5. Epub 2020 Mar 9. PMID 32152808

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04440514/Prot_000.pdf
  • Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04440514/ICF_001.pdf